CLINICAL TRIAL: NCT00001213
Title: Trial of Topical Cysteamine in the Treatment of Corneal Cystine Crystal Accumulation in Cystinosis
Brief Title: Cysteamine Eye Drops to Treat Corneal Crystals in Cystinosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 860062; 86-EI-0062
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Cystinosis
Keywords: Cysteamine Eye Drops; Nephropathic Cystinosis; Corneal Crystals; Benzalkonium; Toxicity; Efficacy; Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteamine topical solution (Experimental): Cysteamine topical solution administered hourly while awake in both eyes
  Interventions: Drug: Cysteamine

INTERVENTIONS:
Drug: Cysteamine

SUMMARY:
Cystinosis is an inherited disease that results in poor growth and kidney disease, among other things. The damage to the kidneys and other organs is thought to be due to accumulation of cystine inside the cells of various body tissues. This chemical also accumulates in the cornea-the covering of the eye over the pupil and iris. After 10 to 20 years, the corneas of some patients become so packed with crystals that the surfaces may become irregular, occasionally causing small, painful breaks.

Patients enrolled in a NIH study on cystinosis are receiving the drug cysteamine. Taken by mouth, this drug reduces cystine in some tissues, but not in the cornea. This study began in 1986 to test whether cysteamine eye drops could prevent or reduce corneal cystine crystals in these patients. The drops have been very effective in removing crystals and reducing pain in patients who take the medication as directed. Patients who do not take the medication as prescribed do not benefit.

After the effectiveness of the drops was proven, the main purpose was modified to continue to evaluate the long-term safety and effectiveness of cysteamine eye drops for treating cystine crystals in the corneas of patients with cystinosis until the drops are approved by the Food and Drug Administration (FDA). When the New Drug Application (NDA) for the Sigma-Tau standard formulation is granted, this protocol will be terminated.

DETAILED DESCRIPTION:
Protocol 86-EI-0062 began as a randomized, double-masked, placebo controlled study to evaluate the efficacy and safety of 0.5% topical cysteamine but was subsequently amended as a natural history protocol. Additional protocols conducted at the National Eye Institute (NEI) at the National Institutes of Health (NIH) began after this protocol and tested various formulations of cysteamine topical solution for efficacy and safety in patients with cystinosis. Subjects from these NIH protocols testing various formulations were ultimately transferred to this natural history protocol for open-label treatment once it was established that the formulation within this study was the most effective. All subjects enrolled in this protocol received the most effective cysteamine topical solution formulation in both eyes. The control was defined as the natural course of corneal crystal accumulation in patients with cystinosis. The efficacy data were obtained from all of the studies conducted at NIH evaluating various cysteamine ophthalmic solution formulations from 1986 until 2005. The safety data were collected from 1986 until the termination of this protocol in July 2013.

OBJECTIVE:

The free thiol cysteamine depletes cystinotic leukocytes and other cells of cystine, whose accumulation is considered the cause of organ damage in cystinosis. This organ damage involves most tissues of the body. Cysteamine therapy improved growth and stabilized renal function in pre-renal transplant cystinosis, without substantial toxicity but there was no noticeable effect on cystine crystal accumulation in the cornea, most likely because of inadequate local cysteamine concentration in the cornea. Previous studies have shown the safety of cysteamine 0.5% topical solution in benzalkonium chloride and its efficacy in resolving the cystine corneal crystals. The main purpose of this protocol is to maintain topical cysteamine treatment in patients with nephropathic cystinosis until the drops are approved by the FDA. When the NDA for the Sigma-Tau standard formulation is granted, the present protocol (86-EI-0062) will be terminated.

STUDY POPULATION:

Up to 350 adults and children over two years old, who have a confirmed diagnosis of cystinosis will be enrolled.

STUDY DESIGN:

This is an open label treatment protocol. Eligible subjects will receive drops of cysteamine 0.5% topical solution in benzalkonium chloride hourly while awake in both eyes. They will undergo an eye examination at their baseline visit. They will take cysteamine eye drops in both eyes every hour during waking hours. They will return to the NIH Clinical Center for a follow-up safety eye examination one year after the baseline visit, and then every two years thereafter until the drug is available commercially.

OUTCOME MEASURES:

The initial pre-specified primary outcome measure was the reduction of cystine corneal crystals. The post-hoc primary outcome measure (after the protocol was modified) was the collection of safety data.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must have a documented clinical diagnosis of cystinosis.
* Patients should be 2 years old or older.

EXCLUSION CRITERIA:

* Inability to travel to NIH for a baseline examination, after 1 year, and every two years thereafter for follow-up
* Inability to cooperate for slit-lamp examination

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 1986-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel J Bishop, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kaiser-Kupfer MI, Fujikawa L, Kuwabara T, Jain S, Gahl WA. Removal of corneal crystals by topical cysteamine in nephropathic cystinosis. N Engl J Med. 1987 Mar 26;316(13):775-9. doi: 10.1056/NEJM198703263161304. PMID 3821824
- [Background] Kaiser-Kupfer MI, Gazzo MA, Datiles MB, Caruso RC, Kuehl EM, Gahl WA. A randomized placebo-controlled trial of cysteamine eye drops in nephropathic cystinosis. Arch Ophthalmol. 1990 May;108(5):689-93. doi: 10.1001/archopht.1990.01070070075038. PMID 2185723
- [Background] Gahl WA. Cystinosis coming of age. Adv Pediatr. 1986;33:95-126. No abstract available. PMID 3541536
- [Background] Gahl WA, Kuehl EM, Iwata F, Lindblad A, Kaiser-Kupfer MI. Corneal crystals in nephropathic cystinosis: natural history and treatment with cysteamine eyedrops. Mol Genet Metab. 2000 Sep-Oct;71(1-2):100-20. doi: 10.1006/mgme.2000.3062. PMID 11001803
- [Background] Iwata F, Kuehl EM, Reed GF, McCain LM, Gahl WA, Kaiser-Kupfer MI. A randomized clinical trial of topical cysteamine disulfide (cystamine) versus free thiol (cysteamine) in the treatment of corneal cystine crystals in cystinosis. Mol Genet Metab. 1998 Aug;64(4):237-42. doi: 10.1006/mgme.1998.2725. PMID 9758713

RESULTS

PARTICIPANT FLOW:
Groups:
- Cysteamine Topical Solution: Cysteamine topical solution administered hourly while awake in both eyes
  Cysteamine
Period: Overall Study
Arm/Group | Cysteamine Topical Solution
Started | 328
Completed | 310
Not Completed | 18
Not completed — Death | 18

BASELINE CHARACTERISTICS:
Arm/Group | Cysteamine Topical Solution
Number analyzed (Participants) | 328
Age, Continuous [Mean (Standard Deviation); unit: years] — Although 328 participants were initially enrolled, the mean and standard deviation were only obtained for 322 participants.
  years | 13.1 (10.04)
Gender [Number; unit: participants] — Gender was captured for 326 out of 328 participants, the gender of two participants is unknown.
  participants
    Female | 153
    Male | 173

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Since efficacy of ophthalmic cysteamine was established and a New Drug Application (NDA) filed, the post-hoc primary outcome measure is the evaluation of safety information. There was no specified time frame for this outcome measure, as safety data was being collected until the drug became available for commercial purchase in May 2013.
Time Frame: Any Time Point up to 27 Years
Measure: Number; unit: participants
Arm/Group | Cysteamine Topical Solution
Number analyzed (Participants) | 328
participants | 257

2. Primary Outcome: Number of Eyes With a Corneal Cystine Crystal Score (CCCS) Response
Description: Response is defined as a decrease from baseline of at least 1 in Corneal Cystine Crystal Score (CCCS) at any time on study when baseline CCCS is greater than or equal to 1, or CCCS does not increase at least 1 at any time on study when baseline CCCS is less than 1.
  The CCCS is based on a library of slit-lamp photographs of corneas with increasing crystal densities (0-3). Slit-lamp photos were to be taken to assess the extent of the corneal crystal accumulation. To minimize bias when assessing the extent of corneal crystal accumulation, photos were centrally graded at the National Eye Institute (NEI) where each photo was graded independently by masked graders. If more than one CCCS was recorded in a given study year, the highest (worst) CCCS value was used for that year.
  The results were obtained from a combined analyses of the NIH cysteamine studies evaluating various cysteamine ophthalmic solution formulations from 1986 through 2005.
Time Frame: Any Time Point Up to 19 Years
Population: One hundred sixty-one (161) participants were analyzed in the pre-specified intent-to-treat population [defined as patients who received study medication (between 1986 and 2005), and had a baseline and a post-baseline CCCS value]. After 2005, all participants enrolled received open-label treatment and only safety data was obtained.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Cysteamine Topical Solution
Number analyzed (Participants) | 161
Number analyzed (eyes) | 321
eyes | 98

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected throughout the study. No specified time period is noted, as participants were followed until the drug became available commercially.
Description: Cystinosis patients typically have multiple medical problems, including kidney failure. The AEs reported do not reflect these systemic problems, focusing instead on ocular AEs (e.g., renal failure is noted in only 2 of 328 patients, though the majority have been managed for kidney disease and/or failure and have received a kidney transplant).
Arm/Group | Cysteamine Topical Solution
Serious Adverse Events (participants affected / at risk) | 11/328
Other Adverse Events (participants affected / at risk) | 257/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysteamine Topical Solution (N=328)
Optic disc disorder (Eye disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Blindness (Eye disorders) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 8 (8)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysteamine Topical Solution (N=328)
Photophobia (Eye disorders) | 239 (239)
Conjunctival hyperaemia (Eye disorders) | 69 (69)
Eye pain (Eye disorders) | 66 (66)
Ocular hyperaemia (Eye disorders) | 52 (52)
Eye irritation (Eye disorders) | 49 (49)
Lacrimation increased (Eye disorders) | 23 (23)
Optic disc disorder (Eye disorders) | 19 (19)
Vision blurred (Eye disorders) | 20 (20)
Keratitis (Eye disorders) | 19 (19)
Dry eye (Eye disorders) | 14 (14)
Eye pruritis (Eye disorders) | 13 (13)
Conjunctivitis (Eye disorders) | 12 (12)
Eyelid oedema (Eye disorders) | 12 (12)
Retinal disorder (Eye disorders) | 11 (11)
Blindness (Eye disorders) | 9 (9)
Corneal epithelium disorder (Eye disorders) | 6 (6)
Blepharitis (Eye disorders) | 5 (5)
Erythema of eyelid (Eye disorders) | 5 (5)
Eye swelling (Eye disorders) | 3 (3)
Conjunctival oedema (Eye disorders) | 2 (2)
Eye oedema (Eye disorders) | 1 (1)
Eyelid cyst (Eye disorders) | 1 (1)
Eyelid irritation (Eye disorders) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 94 (94)
Visual field defect (Nervous system disorders) | 35 (35)
Benign intracranial hypertension (Nervous system disorders) | 4 (4)
Instillation site irritation (General disorders) | 33 (33)
Instillation site pain (General disorders) | 22 (22)
Adverse drug reaction (General disorders) | 7 (7)
Instillation site erythema (General disorders) | 5 (5)
Swelling (General disorders) | 2 (2)
Drug ineffective (Eye disorders) | 1 (1)
Instillation site lacrimation (General disorders) | 1 (1)
Instillation site reaction (General disorders) | 1 (1)
Eye infection (Infections and infestations) | 6 (6)
Conjunctivitis ineffective (Infections and infestations) | 3 (3)
Hordeolum (Infections and infestations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Visual evoked potentials abnormal (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the progressive nature of the drug's development, this protocol reflects the culmination of cysteamine studies performed at NIH. The combined analyses of the data is presented and not the data or analyses of one individual protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No